CLINICAL TRIAL: NCT06389123
Title: A Novel Molecularly Targeted Theranostic Approach Via the αvβ6 Integrin for the Detection and Treatment of Metastatic Carcinomas
Brief Title: Molecularly Targeted Theranostic Approach for the Detection and Treatment of Metastatic Carcinomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Julie L. Sutcliffe, Ph.D, Professor, University of California, Davis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1788760
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Cancer
Keywords: integrin; PET; Theranostics; metastatic cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Single treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [177Lu]Lu DOTA-ABM-5G single dose therapy study (Experimental): Patients will be undergo [68Ga]Ga DOTA-5G PET/CT scans to confirm eligibility for the [177Lu]Lu DOTA-ABM-5G therapy. Patients with sufficient lesion uptake of [68Ga]Ga DOTA-5G PET/CT will be offered therapy.
  Interventions: Drug: [68Ga]Ga DOTA-5G and [177Lu]Lu DOTA-ABM-5G.

INTERVENTIONS:
Drug: [68Ga]Ga DOTA-5G and [177Lu]Lu DOTA-ABM-5G. — Patients will be undergo [68Ga]Ga DOTA-5G PET/CT scans to confirm eligibility for the [177Lu]Lu DOTA-ABM-5G therapy. Patients with sufficient lesion uptake of [68Ga]Ga DOTA-5G PET/CT will be offered therapy. Patients will undergo a follow up [68Ga]Ga DOTA-5G PET/CT scans to assess tretament efficacy.
  Other Names: [68Ga]Ga DOTA-5G; [177Lu]Lu DOTA-ABM-5G; [68Ga]Ga DOTA-5G and [177Lu]Lu DOTA-ABM-5G theranostic pair

SUMMARY:
This is a Phase I study to evaluate the safety and efficacy of the [68Ga]Ga DOTA-5G and [177Lu]Lu DOTA-ABM-5G theranostics pair in patients with metastatic cancer.

DETAILED DESCRIPTION:
This is a Phase I study to evaluate the safety and efficacy of the [68Ga]Ga DOTA-5G and [177Lu]Lu DOTA-ABM-5G theranostics pair in patients with metastatic cancer. [68Ga]Ga DOTA-5G PET/CT will be used to identify and stratify patients eligible for (and most likely to respond to) the [177Lu]Lu DOTA-ABM-5G therapy. Up to 40 patients will be enrolled over a 36-month period with metastatic cancer with a life expectancy of at least 3 months, who demonstrate disease progression after at least 1 prior treatment for metastatic disease and have available archival tissue.

The hypothesis are that a) [68Ga]Ga DOTA-5G will detect lesions in patients with metastatic cancer, b) the theranostic pair [68Ga]Ga DOTA-5G/ [177Lu]Lu DOTA-ABM-5G will be safe and well tolerated, and c) a therapeutic response will be achieved with a single dose of [177Lu]Lu DOTA-ABM-5G.

ELIGIBILITY:
Inclusion Criteria:

[68Ga]Ga DOTA-5G PET/CT Inclusion Criteria:

1. Ability to understand and willingness to sign a written informed consent document.
2. Age 18 or more years
3. Pathologically confirmed GU, GI, breast, cervical, uterine, or head and neck cancers with metastatic disease and measurable disease per RECIST (version 1.1) (i.e. at least 1 lesion > 1 cm or lymph node > 1.5 cm in short axis)
4. Participant must have documented tumor progression for metastatic disease during or following at least one prior FDA approved systemic regimen (Androgen Deprivation allowed) as established by diagnostic imaging.
5. Available archival tumor tissue (excisional, core, or FNA is acceptable). Tissue from a metastatic site is preferred when available.
6. Eastern Cooperative Oncology Group Performance Status ≤ 2
7. Participant must have completed prior systemic therapy at least 2 weeks (washout period) prior to [68Ga]Ga DOTA-5G PET scan. Any clinically significant toxicity (with the exceptions of hair loss and sensory neuropathy) related to prior therapy resolved to Grade 1 or baseline.
8. Hematologic parameters defined as:

Absolute neutrophil count (ANC) ≥ 1000 cells/mm3 Platelet count ≥ 100,000/mm3 Hemoglobin ≥ 8 g/dL

Blood chemistry levels defined as:

AST, ALT, alkaline phosphatase ≤ 5 times upper limit of normal (ULN) Total bilirubin ≤ 2 times ULN Creatinine ≤ 2 times ULN 10. Anticipated life expectancy ≥ 3 months 11. Able to remain motionless for up to 30-60 minutes per scan

[177Lu]Lu DOTA-ABM-5G therapy Inclusion Criteria:

1. Completion of entry into [68Ga]Ga DOTA-5G PET study and completion of scan
2. The presence of at least one measurable disease by [68Ga]Ga DOTA-5G PET/CT (SUVmax>2-fold above normal bone, brain, lung or liver and identified on standard of care diagnostic imaging)

Exclusion Criteria:

[68Ga]Ga DOTA-5G and [177Lu]Lu DOTA-ABM-5G therapy Exclusion Criteria:

1. Participants with Class 3 or 4 NYHA Congestive Heart Failure
2. Clinically significant bleeding within two weeks prior to trial. entry (e.g. gastrointestinal bleeding, intracranial bleeding)
3. Pregnant or lactating women
4. Major surgery, defined as any surgical procedure that involves general anesthesia and a significant incision (i.e., larger than what is required for placement of a central venous access, percutaneous feeding tube, or biopsy) within 28 days prior to study day 1 or anticipated surgery within the subsequent 6 weeks
5. Has an additional active malignancy requiring therapy within the past 2 years (other than early stage, surgically managed basal and squamous skin cancer and in situ malignancies of the breast and cervix)
6. Active, uncontrolled bacterial, viral, or fungal infection(s) despite systemic therapy
7. Psychiatric illness/social situations that would interfere with compliance with study requirements
8. Cannot undergo PET/CT or SPECT/CT scanning because of weight limits (350 lbs.)
9. Pathologically confirmed NSCLC with metastatic disease
10. INR >2.0: PTT>15 seconds above ULN
11. Participant on therapeutic warfarin anticoagulation
12. External beam radiation therapy (EBRT) or radiopharmaceutical treatment within 21 days prior to study day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
[68Ga]Ga DOTA-5G PET/CT imaging | 2 hours from time of injection
  To assess the ability of [68Ga]Ga DOTA-5G to detect lesions in patients with metastatic cancer

SECONDARY OUTCOMES:
[177Lu]Lu DOTA-ABM-5G treatment | 30 days from time of treatment
  To assess the safety and tolerability of a single treatment with [177Lu]Lu DOTA-ABM-5G
[177Lu]Lu DOTA-ABM-5G treatment efficacy | 60 days from time of treatment
  To assess treatment efficacy (response vs. no response) assessed by comparison with a post-treatment scan (standard of care imaging and post second [68Ga]Ga DOTA-5G PET/CT, prior to next line of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Julie L Sutcliffe, Principal Investigator — University of California, Davis
Locations (1):
- The University of California Davis Comprehensive Cancer Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No